CLINICAL TRIAL: NCT05127005
Title: A Multi-center, Investigator-blinded, Randomized, Parallel Group, Superiority Study to Compare the Efficacy of Trapeziectomy Versus Sham Surgery in the Treatment of Osteoarthritis at the Base of the Thumb
Brief Title: Efficacy of Trapeziectomy Versus Sham Surgery in the Treatment of Osteoarthritis at the Base of the Thumb
Acronym: FINTASY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Central Finland Central Hospital (Unknown); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Jarkko Jokihaara, Associate professor, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAUH_FINTASY
Record Dates: First submitted 2021-11-18; First posted 2021-11-19 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Thumb Osteoarthritis
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trapeziectomy (Experimental): Trapeziectomy
  Interventions: Procedure: Trapeziectomy
- Sham surgery (Sham Comparator): Sham surgery
  Interventions: Procedure: Sham
- Non-randomized observational arm (Other): Non-randomized observational arm (trapeziectomy, not blinded)
  Interventions: Procedure: Trapeziectomy

INTERVENTIONS:
Procedure: Trapeziectomy — Surgical excision of trapezoideum
  Arms: Non-randomized observational arm; Trapeziectomy
Procedure: Sham — Skin incision only
  Arms: Sham surgery

SUMMARY:
A multi-center randomized placebo-controlled clinical trial which determines the efficacy of trapeziectomy in patients with persistent painful osteoarthritis at the base of the thumb. The primary outcome is patient reported evaluation of pain and function of the wrist and hand at 6 months after the randomization to treatment group.

DETAILED DESCRIPTION:
A multi-center randomized placebo-controlled clinical trial which determines the efficacy of trapeziectomy in patients with persistent painful osteoarthritis at the base of the thumb (CMC1). The primary outcome is Patient Reported Wrist and Hand Evaluation (PRWHE) at 6 months after the randomization to treatment group. Secondary measures include PRWHE at 3 months, 1 year, 2 years and 5 years, grip strength, and global assessment of change.

ELIGIBILITY:
Inclusion Criteria:

1. Primary thumb basal joint (CMC1) osteoarthritis (Eaton Glickel grade 2 or higher) confirmed by standard x-rays and with symptoms limiting activities of daily living
2. Indication for surgical treatment of thumb basal joint (CMC1) osteoarthritis after insufficient benefit from non-operative treatment, including use of a thumb orthosis and pain medication (NSAIDs or paracetamol, implemented for at least three months.
3. Thumb pain in use of at least 4 on a 0 to10 numerical rating scale (NRS, 10=worst pain)
4. Age > 45 years
5. ASA-classification I-II (American Society for Anesthesiologist's Physical Status Classification System)
6. Ability to speak, understand and read in the language of the clinical site
7. Provision of informed consent from the participant

Exclusion Criteria:

1. Patients' main complaint is due to some other problem than primary thumb basal joint (CMC1) osteoarthritis or patient will undergo any other surgery in conjunction with trapeziectomy
2. Neurologic condition affecting the function or symptoms of the upper extremity
3. <6 months from other surgical procedure of the upper extremities
4. Rheumatoid arthritis or other inflammatory joint disease
5. Bilateral thumb basal joint (CMC1) osteoarthritis in which patient requests treatment for both sides
6. Previous operation due tothumb basal joint (CMC1) osteoarthritis for either side
7. >45 degrees of hyperextension in the thumb MP joint in resting position (zig zag deformity)
8. Patient is unable to continue his/her current job due to thumb pain

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Patient reported wrist and hand evaluation (PRWHE) | 6 months
  PROM questionnaire

SECONDARY OUTCOMES:
Patient reported wrist and hand evaluation (PRWHE) | 3 months, and 1, 2, 5 years
  PROM questionnaire
Global improvement | 3 and 6 months, and 1, 2, and 5 years
  PROM, question (Likert scale)
Patient accepted symptom state | 3 and 6 months, and 1, 2, and 5 years
  PROM, question (Likert scale)
Grip and pinch strength | 6 months
  Measured with dynamometer
EUROQOL EQ-5D-5L | 3 and 6 months, and 1, 2, and 5 years
  PROM, health-related quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jarkko Jokihaara, Study Chair — TAUH
Locations (4):
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No
In this trial IPD sharing is restricted by data protection regulations